CLINICAL TRIAL: NCT07277088
Title: A Prospective, Single-center, Randomized Controlled Clinical Study to Evaluate the Efficacy and Safety of the Percutaneous Interventional Surgery Control System for Pulmonary Nodule Biopsy
Brief Title: The Percutaneous Interventional Surgery Control System for Pulmonary Nodule Biopsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiayuan Sun (Other)
Collaborators: Shanghai United Imaging Intelligence Co., Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Chief Physician, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IS25177
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Nodules; Lung Cancer (Diagnosis); Percutaneous Needle Biopsy; Transthoracic Needle Biopsy; Robotic Assisted Intervention
Keywords: Percutaneous Needle Biopsy; Transthoracic Needle Biopsy; Pulmonary Nodules; Lung Cancer (Diagnosis); Robotic Assisted Intervention
MeSH Terms: conditions — Multiple Pulmonary Nodules; Lung Neoplasms; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic assisted group (Experimental): Patients undergo percutaneous needle biopsy of pulmonary nodules assisted by a percutaneous interventional surgical control system. The system performs automatically needle positioning and puncture.
  Interventions: Diagnostic Test: Percutaneous Needle Biopsy with Interventional Surgical Control System
- Manual group (Active Comparator): Patients receive traditional manual percutaneous needle biopsy of pulmonary nodules, operated by experienced interventional physicians.
  Interventions: Diagnostic Test: Conventional Manual Percutaneous Needle Biopsy

INTERVENTIONS:
Diagnostic Test: Percutaneous Needle Biopsy with Interventional Surgical Control System — Patients undergo percutaneous needle biopsy of pulmonary nodules with assistance from a percutaneous interventional surgical control system. The system performs automatically needle positioning and puncture.
  Other Names: Robotic assisted PTNB
  Arms: Robotic assisted group
Diagnostic Test: Conventional Manual Percutaneous Needle Biopsy — Patients receive traditional manual percutaneous needle biopsy of pulmonary nodules under CT guidance, operated by experienced interventional physicians.
  Other Names: Conventional PTNB
  Arms: Manual group

SUMMARY:
This prospective, single-center, non-inferiority, randomized controlled clinical trial aims to evaluate the efficacy and safety of a percutaneous interventional surgical control system in performing percutaneous needle biopsy of pulmonary nodules, compared with conventional manual biopsy. The study will be conducted at Shanghai Chest Hospital and plans to enroll 158 patients who meet the indications for percutaneous transthoracic needle biopsy (PTNB) and have no contraindications. Participants will be randomly assigned to one of two groups: the experimental group will undergo PTNB assisted by the percutaneous interventional surgical control system, while the control group will receive traditional manual PTNB. The primary endpoint is diagnostic yield; secondary endpoints include technical success rate, number of needle adjustments, puncture time, total procedure time, radiation dose, and complication rates.

ELIGIBILITY:
Inclusion Criteria:

1) Age ranging from 18 years old to 80 years old, gender not restricted; 2) Patients with pulmonary nodules detected by chest CT, suspected to be malignant and judged by the researchers to require puncture biopsy for a clear diagnosis; 3) Pulmonary nodules with a long diameter greater than 8mm but not exceeding 30mm; 4) Have signed the informed consent form and voluntarily participate in this clinical study; 5) Can understand this research and cooperate with the research procedures, and can follow the requirements for follow-up observation.

Exclusion Criteria:

1) Subjects with irreparable coagulation dysfunction, infectious lesions on the puncture path, lesions adjacent to organs or surrounded by large blood vessels, suspected pulmonary echinococcosis on imaging, patients on mechanical ventilation (with a ventilator), liver multilocular echinococcosis, coma or other patients who are uncooperative; 2) Those judged by the investigators to be unsuitable for chest percutaneous puncture surgery: such as severe pulmonary hypertension, pulmonary bullae, chronic obstructive pulmonary disease, emphysema, pulmonary fibrosis; 3) Poor overall condition (multiple systemic metastases, severe infection, high fever), obvious cachexia, severe dysfunction of important organs, severe anemia and nutritional metabolic disorders that cannot be improved in the short term; 4) Those allergic to contrast agents or anesthetics; 5) Implantation of pacemakers; 6) Pregnant or lactating women, or those with a fertility plan during the clinical trial; 7) Patients who cannot cooperate with the doctor to complete the puncture surgery, such as known drug or alcohol addiction, mental and neurological diseases, intellectual disability, psychological disorders, etc.; 8) Those participating in another drug or medical device clinical trial (within 3 months of drug clinical trial or within 1 month of medical device clinical trial); 9) The target lesion has been diagnosed or has received treatment; 10) Other situations that the investigator deems not suitable for this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Dianostic yield | Up to 6 months after biopsy
  Malignant lesions and specific benign lesions (e.g., fungal infections, tuberculosis, granulomas, etc.) are considered as having a definitive diagnosis.
  Non-specific benign lesions (e.g., inflammation) are deemed diagnosed if they are confirmed by at least 6 months of follow-up, surgical resection, other biopsy methods, or radiological follow-up showing lesion shrinkage or disappearance.
  Atypical cells or normal lung tissue are classified as non-diagnostic.

SECONDARY OUTCOMES:
Technical Success Rate | Intra-operative
  Defined as the successful positioning of the biopsy needle to the target lesion by the investigator based on intra-operative CT, without the use of other auxiliary puncture tools or needle guidance techniques. If yes, it is defined as technically successful. Technical success rate = (Number of patients with technical success / Total number of participants) × 100%.
Number of Needle Adjustments | Intra-operative
  The number of needle adjustments from the moment the first needle tip touches the skin until the researcher confirms the puncture is successful, recorded by the investigator during the procedure. Any change in puncture direction, needle withdrawal, or needle removal after needle insertion should be counted.
Puncture time | Intra-operative
  Refers to the duration from when the needle tip first reaches the skin puncture site to when successful puncture is confirmed (i.e., when the investigator judges that biopsy can be performed based on intra-operative CT scan).
Procedural Time | Intra-operative
  Refers to the total time from when the patient is positioned to when the procedure is completed.
Complication rate | Up to 6 months after biopsy
  Common complications of percutaneous needle biopsy include puncture site infection, pneumothorax, bleeding, hemoptysis, pleural reaction, etc. Rare complications include air embolism, cardiac tamponade, tumor seeding along the needle tract, nerve injury, etc.
Radiation dose | Intra-operative
  The radiation dose received by the patient as recorded by the CT scan protocol during the biopsy procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anzidei M, Argiro R, Porfiri A, Boni F, Anile M, Zaccagna F, Vitolo D, Saba L, Napoli A, Leonardi A, Longo F, Venuta F, Bezzi M, Catalano C. Preliminary clinical experience with a dedicated interventional robotic system for CT-guided biopsies of lung lesions: a comparison with the conventional manual technique. Eur Radiol. 2015 May;25(5):1310-6. doi: 10.1007/s00330-014-3508-z. Epub 2014 Nov 23. PMID 25417130
- [Result] Appelbaum L, Sosna J, Nissenbaum Y, Benshtein A, Goldberg SN. Electromagnetic navigation system for CT-guided biopsy of small lesions. AJR Am J Roentgenol. 2011 May;196(5):1194-200. doi: 10.2214/AJR.10.5151. PMID 21512092
- [Result] Alexander ES, Petre EN, Bodard S, Marinelli B, Sarkar D, Cornelis FH. Comparison of a Patient-Mounted Needle-Driving Robotic System versus Single-Rotation CT Fluoroscopy to Perform CT-Guided Percutaneous Lung Biopsies. J Vasc Interv Radiol. 2024 Jun;35(6):859-864. doi: 10.1016/j.jvir.2024.02.023. Epub 2024 Mar 5. PMID 38447771
- [Result] Lee KH, Lim KY, Suh YJ, Hur J, Han DH, Kang MJ, Choo JY, Kim C, Kim JI, Yoon SH, Lee W, Park CM. Diagnostic Accuracy of Percutaneous Transthoracic Needle Lung Biopsies: A Multicenter Study. Korean J Radiol. 2019 Aug;20(8):1300-1310. doi: 10.3348/kjr.2019.0189. PMID 31339018
- [Result] Rivera MP, Mehta AC, Wahidi MM. Establishing the diagnosis of lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e142S-e165S. doi: 10.1378/chest.12-2353. PMID 23649436
- [Result] Chang YY, Chen CK, Yeh YC, Wu MH. Diagnostic feasibility and safety of CT-guided core biopsy for lung nodules less than or equal to 8 mm: A single-institution experience. Eur Radiol. 2018 Feb;28(2):796-806. doi: 10.1007/s00330-017-5027-1. Epub 2017 Sep 7. PMID 28884222
- [Result] Horeweg N, van Rosmalen J, Heuvelmans MA, van der Aalst CM, Vliegenthart R, Scholten ET, ten Haaf K, Nackaerts K, Lammers JW, Weenink C, Groen HJ, van Ooijen P, de Jong PA, de Bock GH, Mali W, de Koning HJ, Oudkerk M. Lung cancer probability in patients with CT-detected pulmonary nodules: a prespecified analysis of data from the NELSON trial of low-dose CT screening. Lancet Oncol. 2014 Nov;15(12):1332-41. doi: 10.1016/S1470-2045(14)70389-4. Epub 2014 Oct 1. PMID 25282285
- [Result] Baldwin DR, Callister ME; Guideline Development Group. The British Thoracic Society guidelines on the investigation and management of pulmonary nodules. Thorax. 2015 Aug;70(8):794-8. doi: 10.1136/thoraxjnl-2015-207221. Epub 2015 Jul 1. PMID 26135833
- [Result] Han B, Zheng R, Zeng H, Wang S, Sun K, Chen R, Li L, Wei W, He J. Cancer incidence and mortality in China, 2022. J Natl Cancer Cent. 2024 Feb 2;4(1):47-53. doi: 10.1016/j.jncc.2024.01.006. eCollection 2024 Mar. PMID 39036382